CLINICAL TRIAL: NCT02957136
Title: Randomized Clinical Trial of Multi-respiratory Pathogen Testing Versus Usual Care in Emergency Department (ED) Patients With Upper Respiratory Symptoms
Brief Title: Rapid Diagnostics for Upper Respiratory Infections in the Emergency Department
Acronym: URIDxED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: BioFire Diagnostics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 894097
Record Dates: First submitted 2016-10-31; First posted 2016-11-07 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Respiratory Tract Infections; Influenza, Human; Common Cold
Keywords: Respiratory Tract Infections; Influenza, Human; Common Cold; Viral Infection; Pathology, Molecular; Molecular Diagnostics; Diagnostic Testing; Clinical Microbiology; Polymerase Chain Reaction; Antibiotic Stewardship; Antimicrobial Use; Emergency Department; Emergency Room
MeSH Terms: conditions — Respiratory Tract Infections; Influenza, Human; Common Cold; Virus Diseases; Emergencies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rapid respiratory pathogen test arm (Experimental): ED patients in this arm will receive a rapid respiratory pathogen nucleic acid amplification test plus usual care.
  Interventions: Device: Rapid respiratory pathogen nucleic acid amplification test
- Usual care control arm (No Intervention): ED patients in this arm will receive clinician-directed standard of care, which may include but is not limited to no testing, point-of-care influenza testing, or delayed testing for respiratory pathogens at off-site laboratory.

INTERVENTIONS:
Device: Rapid respiratory pathogen nucleic acid amplification test — Patients randomized to the rapid respiratory pathogen nucleic acid amplification test (Film Array Respiratory Panel, BioFire Diagnostics), will receive usual physician-directed care plus results from a rapid diagnostic test for 20 common respiratory pathogens. Patients will have a nasopharyngeal swab sample collected and tested during the ED episode of care with results reported in the electronic medical record (EMR) within two hours of sample collection. ED physicians will receive education regarding the rapid respiratory pathogen test prior to commencing the study. During the study, ED physicians will be free to review and interpret the respiratory pathogen test results and make treatment decisions based on their individual clinical judgment without involvement of study personnel.
  Arms: Rapid respiratory pathogen test arm

SUMMARY:
This is a randomized clinical trial to assess the effect of rapid, near point-of-care testing for multiple common respiratory viruses and bacteria on antibiotic and anti-influenza medication use in emergency department (ED) patients with symptoms of influenza-like illness (ILI) and/or upper respiratory infection (URI).

DETAILED DESCRIPTION:
This is a randomized clinical trial to assess the effect of rapid, near point-of-care testing for multiple common respiratory viruses and bacteria on antibiotic and anti-influenza medication use in emergency department (ED) patients with symptoms of influenza-like illness (ILI) and/or upper respiratory infection (URI). The intervention is a rapid, multi-respiratory pathogen nucleic acid amplification panel test (FilmArray Respiratory Panel; BioFire Diagnostics, LLC) with clinical result reporting within two hours of sample collection. Randomization is at the individual patient level. Intervention patients will receive usual care plus the rapid multi-respiratory pathogen test. Control patients will receive physician-directed usual care without the rapid, multi-respiratory pathogen test, which may include but is not limited to no testing, point-of-care influenza testing, or delayed testing for multiple respiratory pathogens at an off-site laboratory. The primary outcome is antibiotic administration or prescription during the initial ED episode of care. The investigators primary hypothesis is that rapid multi-respiratory pathogen testing will be associated with a ≥15% reduction in antibiotic use in intervention patients, relative to control patients (usual care). The investigators secondary outcome is administration or prescription of antivirals during the initial ED episode of care. The investigators secondary hypothesis is that rapid multi-respiratory pathogen testing will improve anti-influenza medication use in intervention patients (composite rate of anti-influenza treatment in positive patients and non-use of anti-influenza treatment in negative patients), relative to control patients receiving usual care alone.

ELIGIBILITY:
Inclusion Criteria:

* University of California, Davis (UC Davis) Emergency Department patients evaluated for influenza like illness and/or upper respiratory infection by an ED physician who consent and agree to have a nasopharyngeal swab collected for the study
* English speaking or Spanish speaking patients

Exclusion Criteria:

* Neonates
* Prisoners
* Employees of UC Davis/Students of the Principal Investigator or Co-Principal Investigator
* Non-English, non-Spanish speaking patients

Ages: 1 Year to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2016-12-08 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Polage, MD, MAS, Principal Investigator — Duke University; Larissa May, MD, MSPH, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] May L, Tatro G, Poltavskiy E, Mooso B, Hon S, Bang H, Polage C. Rapid Multiplex Testing for Upper Respiratory Pathogens in the Emergency Department: A Randomized Controlled Trial. Open Forum Infect Dis. 2019 Nov 5;6(12):ofz481. doi: 10.1093/ofid/ofz481. eCollection 2019 Dec. PMID 32128326

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from rapid care and main adult and pediatric ED areas between December 2016 and April 2018.
Period: Overall Study
Arm/Group | Rapid Respiratory Pathogen Test Arm | Usual Care Control Arm
Started | 95 | 99
Completed | 93 | 98
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rapid Respiratory Pathogen Test Arm | Usual Care Control Arm | Total
Number analyzed (Participants) | 93 | 98 | 191
Age, Customized [Count of Participants; unit: Participants]
  Pediatric (1-17 y) | 32 | 39 | 71
  Adults (18 y or older) | 61 | 59 | 120
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 55 | 110
  Male | 38 | 43 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 32 | 59
  Not Hispanic or Latino | 66 | 66 | 132
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 1 | 6
  Asian | 3 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 18 | 17 | 35
  White | 43 | 44 | 87
  More than one race | 20 | 29 | 49
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 93 | 98 | 191

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Receiving Antibiotics or a Prescription for Antibiotics in the ED
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Rapid Respiratory Pathogen Test Arm | Usual Care Control Arm
Number analyzed (Participants) | 93 | 98
Participants | 20 | 33

2. Secondary Outcome: Proportion of Patients With a Respiratory Pathogen Identified
Description: Any respiratory pathogen detected by the FilmArray Respiratory Panel test or other diagnostic test ordered by the physician
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Rapid Respiratory Pathogen Test Arm | Usual Care Control Arm
Number analyzed (Participants) | 93 | 98
Participants | 61 | 20

3. Secondary Outcome: Proportion of Patients With a Laboratory-confirmed Influenza Diagnosis
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Rapid Respiratory Pathogen Test Arm | Usual Care Control Arm
Number analyzed (Participants) | 93 | 98
Participants | 24 | 8

4. Secondary Outcome: Proportion of Patients Receiving Appropriate Anti-influenza Treatment or Prescription
Description: Composite rate of anti-influenza treatment in positive patients and non-use of anti-influenza treatment in negative patients
Time Frame: Day 0
Population: Analysis limited to population receiving an Influenza test defining positive or negative laboratory confirmed Influenza status.
Measure: Count of Participants; unit: Participants
Arm/Group | Rapid Respiratory Pathogen Test Arm | Usual Care Control Arm
Number analyzed (Participants) | 93 | 37
Participants | 73 | 32

5. Secondary Outcome: Proportion of Patients Discharged Home From the ED Versus Hospital Admission
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Rapid Respiratory Pathogen Test Arm | Usual Care Control Arm
Number analyzed (Participants) | 93 | 98
Participants | 69 | 66

6. Secondary Outcome: Proportion of Patients With All-cause or Respiratory Illness-related Repeat ED Visit, Hospital or ICU Admission, or Death Within 30 Days
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Rapid Respiratory Pathogen Test Arm | Usual Care Control Arm
Number analyzed (Participants) | 93 | 98
Participants | 31 | 38

7. Secondary Outcome: Proportion of of Patients With Clinician Adherence to Guidelines for the Treatment of Patients With Influenza (Recommendations for Use of Antivirals Only)
Time Frame: Day 0
Population: Analysis limited to patients with influenza test and positive influenza result.
Measure: Count of Participants; unit: Participants
Arm/Group | Rapid Respiratory Pathogen Test Arm | Usual Care Control Arm
Number analyzed (Participants) | 24 | 8
Participants | 7 | 3

8. Secondary Outcome: Median Length of ED Stay
Time Frame: Day 0
Measure: Median (Full Range); unit: hours
Arm/Group | Rapid Respiratory Pathogen Test Arm | Usual Care Control Arm
Number analyzed (Participants) | 93 | 98
hours | 4.7 [1.5 to 15.2] | 5.0 [1.6 to 13.1]

9. Secondary Outcome: Median Length of Hospital Stay
Time Frame: 30 days
Measure: Median (Full Range); unit: hours
Arm/Group | Rapid Respiratory Pathogen Test Arm | Usual Care Control Arm
Number analyzed (Participants) | 20 | 27
hours | 71.2 [23.8 to 441] | 54.93 [5.4 to 343]

ADVERSE EVENTS:
Time Frame: 30 days
Description: Collected all-cause mortality at 30 days, hospitalization (disposition from initial ED study visit), 30-day revisit to ED (all, respiratory illness-related, nonrespiratory illness related)
Arm/Group | Rapid Respiratory Pathogen Test Arm | Usual Care Control Arm
All-Cause Mortality (participants affected / at risk) | 1/93 | 0/98
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/98
Other Adverse Events (participants affected / at risk) | 0/93 | 0/98

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT02957136/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT02957136/ICF_001.pdf